CLINICAL TRIAL: NCT05351528
Title: Relationship Between Burdens and Healthy Lifestyle Behaviors of Caregiver Family Members for the Disabled in Bukhara
Brief Title: of Caregiver Family Members for the Disabled in Bukhara
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Nurhayat KORKMAZ, Principal Investigator, Karadeniz Technical University
Other Study IDs: KTU-SBU-FTR-01
Record Dates: First submitted 2022-04-11; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Caregiver Burden
Keywords: handicapped; caregiver burden; healthy lifestyle
MeSH Terms: conditions — Caregiver Burden | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Caregiver burden and healthy lifestyle behaviors were evaluated.

SUMMARY:
The responsibilities of caring for a disabled family member may cause caregivers to develop risky behaviors for caregiver's health. Therefore, we aimed to examine the relationship between caregiver burdens and healthy lifestyle behaviors of family members caring for a disabled child.

DETAILED DESCRIPTION:
In the study, family members living in Bukhara, Uzbekistan, and caring for a disabled person under the age of 24 were evaluated. Caregiver burden was evaluated with the Caregiver Burden Scale and healthy lifestyle behaviors were evaluated with the Healthy Lifestyle Behaviors Scale II. The fact that there is no earlier study on caregivers of disabled people in Uzbekistan and no research in the literature examining the relationship between caregiving burden and healthy lifestyle behaviors in individuals with disabled children, make this study unique.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Having a disabled child to take care of
* Being literate

Exclusion Criteria:

* The age of the disabled person being cared for is over 24 years old.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Caregiver Family Member with disabled children
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Socio-demographic information | Two months
  Age, height, body weight, employment status, income status, marital status
Number of child | Two months
  Number of healthy and disabled children
Assessment of the child age | Two months
  Age
Assessment of the child | Two months
  Gender
Caregiver Burden Scale | Two months
  The scale has a Likert-type rating ranging from 0 to 4 as "never, rarely, sometimes, quite often, almost always". A minimum of 0 and a maximum of 88 points can be obtained from the scale. The items in the scale are generally related to the social and emotional domain, and a high score indicates a high level of distress.

SECONDARY OUTCOMES:
Healthy Lifestyle Behaviors Scale II | Two months
  The scale is scored as "never (1)-regularly (4)". The lowest score for the whole scale is 52 and the highest score is 208. The high scores obtained from the scale indicate how high the individual applies the specified health behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Nurhayat Korkmaz, PhDstudent, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No